CLINICAL TRIAL: NCT06159062
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 162 With a Single Ascending Dose in Subjects With Chronic Hepatitis B Virus Infection
Brief Title: A Clinical Study of 162 in Subjects With Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment difficulty
Sponsor: Yangshengtang Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YST-162-102
Record Dates: First submitted 2023-11-20; First posted 2023-12-06 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 162 (Experimental): The dose-escalation stage will be conducted sequentially at 3 dose cohorts, which are 50 mg in the pre-test, 75 mg and 100 mg in the formal test.
  Two subjects with chronic HBV infection will be enrolled in the 50 mg dose cohort and all will be given the investigational product 162.
  Four subjects with chronic HBV infection will be enrolled in the 75 mg and 100 mg dose cohorts, respectively. Subjects in each cohort will be randomized 3:1 to receive a single ascending dose of investigational product 162 or placebo.
  Interventions: Drug: 162
- Placebo (Placebo Comparator): The dose-escalation stage will be conducted sequentially at 3 dose cohorts, which are 50 mg in the pre-test, 75 mg and 100 mg in the formal test.
  Two subjects with chronic HBV infection will be enrolled in the 50 mg dose cohort and all will be given the investigational product 162.
  Four subjects with chronic HBV infection will be enrolled in the 75 mg and 100 mg dose cohorts, respectively. Subjects in each cohort will be randomized 3:1 to receive a single ascending dose of investigational product 162 or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 162 — The investigational product 162 is a novel monoclonal antibody targeting HBsAg.
  Arms: 162
Drug: Placebo — Placebo do not consist any active ingredients.
  Arms: Placebo

SUMMARY:
The goal of this intervention research is to learn about the safety and tolerability of 162 with a single ascending dose in subjects with chronic hepatitis B virus (HBV) infection.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind and placebo-controlled dose escalation study design.

The dose-escalation stage will be conducted sequentially at 3 dose cohorts, which are 50 mg in the pre-test, 75 mg and 100 mg in the formal test.

Two subjects with chronic HBV infection will be enrolled in the 50 mg dose cohort and all will be given the investigational product 162.

Four subjects with chronic HBV infection will be enrolled in the 75 mg and 100 mg dose cohorts, respectively. Subjects in each cohort will be randomized 3:1 to receive a single ascending dose of 162 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able and willing to provide written informed consent and to comply with the study protocol according to ICH and local regulations.

  2. Positive serum HBsAg and/or HBV DNA status for > 6 months prior to screening (two documented positive HBsAg and/or HBV DNA tests at least 6 months apart, one of which is at screening) or previous liver biopsy results with chronic HBV infection.

  3. On Nucleos(t)ide analogs therapy for at least 3 months without an interruption of 7 or more consecutive days before the screening, and expected to remain on the same Nucleos(t)ide analogs for the duration of study participation.

  4. 500 ≤ HBsAg ≤ 3,000 IU/mL, HBV DNA ≤ 20 IU/mL and ALT ≤ 3×ULN. 5. A male subject must agree to use adequate contraception from screening through at least 24 weeks after the dose of investigational product. Refer to Section 5.5 for more information on highly effective methods of contraception.

  6. Women of childbearing potential must have a negative pregnancy test prior to the dosing administration, and agree to use adequate contraception from screening through at least 24 weeks after the dose of investigational product. A female subject of non-childbearing potential will have had at least 12 continuous months of natural (spontaneous) amenorrhoea, follicle stimulating hormone (FSH) level > 40 mIU/mL at screening, and an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms); or have had surgical bilateral oophorectomy, hysterectomy or bilateral tubal ligation beyond 6 weeks prior to screening. Refer to Section 5.5 for more information on highly effective methods of contraception.

Exclusion Criteria:

* 1. Patients who had history of anaphylaxis against the active ingredients or excipients of the investigational product 162.

  2. History of allergic reactions to monoclonal antibodies or antibody fragments.

  3. History or presence of clinical significant liver disease other than chronic HBV infection (e.g., autoimmune hepatitis, alcoholic liver disease, non-alcoholic steatohepatitis).

  4. Patients who have impaired cardiac function or clinically significant cardiac diseases, including any of the following: New York Heart Association class III-IV for cardiac insufficiency； Patients with poorly controlled arrhythmia: QTc interval > 480 ms calculated by Fridericia's formula, or congenital syndrome of prolonged QT interval; Any of the following within 6 months prior to the screening: myocardial infarction, severe or unstable angina, congestive heart failure, cerebrovascular accident (including transient ischemic attack), symptomatic pulmonary embolism or other clinically significant thromboembolic disease, or coronary artery bypass graft; Patients with other clinically significant cardiovascular disease who were assessed as unsuitable for this study by the investigator.

  5. Patients with uncontrolled hypertension (systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg) or previous hypertensive crisis or hypertensive encephalopathy.

  6. Patients with other active infections other than HBV infection requiring continual treatment with antibiotics or antivirals (except for clinically insignificant temporary infection such as cold), or positive for hepatitis C virus (HCV) or human immunodeficiency virus (HIV) antibodies at screening.

  7. Patients with history of hepatitis A virus (HAV), hepatitis D virus (HDV) or hepatitis E virus (HEV).

  8. Patients with history of malignant tumor within 5 years except cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of uterine cervix.

  9. History or presence of immune-mediated diseases, including but not limited to idiopathic thrombocytopenic purpura, systemic lupus erythematosus, rheumatoid arthritis.

  10. Liver biopsy, Fibroscan or equivalent test obtained within the past 6 months demonstrating liver with evidence of progressive fibrosis or cirrhosis ( Metavir 3, recommended cut-off for fibroscan 8.5 kPa).

  11. Evidence of liver cirrhosis or decompensated liver disease such as Child-Pugh Class B or C, ascites, esophageal or gastric varices, hepatic encephalopathy or portal hypertension.

  12. History of or suspicion of hepatocellular carcinoma or alpha fetoprotein (AFP) > 50 ng/mL at screening.

  13. History of allogenic transplantation of organs, bone marrow or stem cell. 14. Any other concomitant disease, condition or treatment that could interfere with the conduct of the study or that would, in the opinion of the Investigator or Sponsor, pose an unacceptable risk to the subject in the study or interfere with the interpretation of study data.

  15. Those who received blood transfusion, albumin, recombinant human thrombopoietin, or colony-stimulating factor therapy within 2 weeks prior to screening 16. Patients who have not sufficient baseline organ function and whose laboratory data meet the following criteria at enrollment: Absolute neutrophil count (ANC) < 2.0×109/L; Serum albumin < 35 g/L; Total bilirubin > 1.5×ULN; International normalized ratio (INR) > 1×ULN; Hemoglobin < 100 g/L; Platelets < 80×109/L; Creatinine clearance < 50 mL/min. 17. Patients who had received an immunosuppressant, immunity-modifying drug (e.g., interferon, thymosin agents), cytotoxic chemotherapy that can affect their immune system, or radiation therapy within 6 months prior to the dosing of investigational product, except for the following treatments: a) topical or inhaled corticosteroids; b) short-term (treatment duration up to 7 days) use of systemic glucocorticoids for prevention or treatment of non-autoimmune allergic diseases.

  18. Those who have received live or attenuated vaccines (e.g., measles, mumps, rubella, varicella, yellow fever, rabies, BCG, typhoid vaccine, etc.) within 4 weeks before screening, or any covid-19 vaccine within 2 weeks before screening.

  19. Those who underwent major surgery within 4 weeks before screening, or plan to undergo major surgery during the study.

  20. Those who are participating in other clinical studies, or currently not participating in a study and have been dosed in another clinical study 4 weeks prior to screening, or previous treatment with an investigational agent for chronic HBV infection 6 months prior to screening.

  21. Pregnant or lactating women. 22. Those who are determined disqualified to join clinical studies by investigator for other causes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Adverse event (consists of dose limited toxicity) | From the participant receives the investigational product to 28 days after the investigational product administered
  incidence and severity of adverse events

SECONDARY OUTCOMES:
Area under the concentration curve | Within 30 minutes before the dosing administration to 648 hours after the start of the dosing administration
  Area under the concentration curve
Maximum concentration | Within 30 minutes before the dosing administration to 648 hours after the start of the dosing administration
  Maximum plasma concentration of 162
Half-life | Within 30 min before the dosing administration to 648 h after the start of the dosing administration
  Half-life fo 162 eliminates from plasma
Time of maximum concentration | Within 30 minutes before the dosing administration to 648 hours after the start of the dosing administration
  Time of maximum concentration of 162 in plasma
Concentration of serum Hepatitis B surface antigen (HBsAg) | Within 30 minutes before the dosing administration to 648 hours after the start of the dosing administration
  The concentration of serum Hepatitis B surface antigen (HBsAg)
Concentration of serum Hepatitis B virus DNA | Within 30 minutes before the dosing administration to 648 hours after the start of the dosing administration
  The concentration of serum Hepatitis B virus DNA

CONTACTS AND LOCATIONS:
Locations (1):
- Emeritus Research, Melbourne, Camberwell, Australia

IPD SHARING:
Plan to Share IPD: No